CLINICAL TRIAL: NCT00514293
Title: Phase II Trial of Bexarotene (Targretin) Capsules With Tretinoin and Chemotherapy in Patients With Advanced Non-small-cell Lung Cancer
Brief Title: Bexarotene, Tretinoin, and Combination Chemotherapy in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Raghu Nandan, M.D., Inc (Other)
Responsible Party: Raghu Nandan, R. Nandan M.D. Incorporated
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000561066; EISAI-2007-01-22
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2008-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bexarotene; Capecitabine; Carboplatin; Cisplatin; Docetaxel; Tretinoin

INTERVENTIONS:
Drug: bexarotene
Drug: capecitabine
Drug: carboplatin
Drug: cisplatin
Drug: docetaxel
Drug: tretinoin

SUMMARY:
RATIONALE: Bexarotene and tretinoin may cause tumor cells to look more like normal cells, and to grow and spread more slowly. Drugs used in chemotherapy, such as cisplatin, carboplatin, docetaxel, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bexarotene and tretinoin together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving bexarotene together with tretinoin and combination chemotherapy works in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of bexarotene at a dose of 375 mg daily for 4 days with tretinoin also for the same 3 days with chemotherapy in patients with advanced non-small cell lung cancer.
* Evaluate the safety and tolerability of this drug combination.

OUTLINE: Patients will receive oral bexarotene 375 mg once daily and oral tretinoin 50 mg twice daily on days 1-3. Patients also receive combination chemotherapy comprising cisplatin or carboplatin with docetaxel and capecitabine orally or intravenously on days 1-3. Treatment repeats every 14 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients will be followed every 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIB disease with a malignant pleural effusion
  * Stage IV disease
* Chemotherapy-naive disease
* Brain metastases allowed provided patients have completed radiation treatment with no actively progressing brain metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* Absence of hepatic dysfunction that is characterized by the following:

  * AST/ALT > 3 times upper limit of normal (ULN) (unless due to liver metastases)
  * Bilirubin > 3 times ULN (unless due to liver metastases)
* ANC ≥ 1,500/mm^3
* Platelets ≥ 100,000/mm^3
* Negative pregnancy test prior to the initiation of treatment
* Female and male patients of childbearing potential must agree to sexual abstinence for at least 4 weeks prior to study OR practice 2 reliable forms of effective contraception simultaneously (strongly recommended that one of the two forms of contraception be non-hormonal) at least 4 weeks prior to, during the entire study treatment, and for at least 1 month after treatment is discontinued
* Male patients with female sexual partners who are pregnant, possibly pregnant, or who could become pregnant during the study must agree to use condoms during sexual intercourse during the entire study treatment and for at least 1 month after the last dose of bexarotene
* Must be willing and able to give informed consent, comply with study instructions, and commit to all study visits

Exclusion criteria:

* Pregnancy, intent to become pregnant, or breast-feeding
* Significant concurrent or intercurrent illness
* Risk factor for pancreatitis (e.g., uncontrolled hyperlipidemia, excessive alcohol consumption, uncontrolled diabetes mellitus, biliary tract disease)
* Untreated hypothyroidism
* Active second malignancy with the exception of carcinoma in situ, early-stage prostate cancer, and squamous or basal cell carcinoma of skin
* Unwillingness or inability to minimize exposure to sunlight and artificial ultraviolet light while receiving bexarotene
* Known contraindication (according to product labeling) to Lipitor^® (or another selected lipid lowering agent) or levothyroxine
* Known hypersensitivity to bexarotene or other component of bexarotene

PRIOR CONCURRENT THERAPY:

Inclusion criteria

* Tyrosine kinase inhibitor therapy such as erlotinib hydrochloride is allowed for up to 3 months prior to initiation of this regimen provided the disease is unresponsive to such treatment
* Concurrent radiation therapy administered for symptom relief
* Also see Disease Characteristics

Exclusion criteria

* Prior therapy, except radiation to the brain for palliation, as long as a measurable lesion is still present
* Prior use of bexarotene
* Prior systemic anticancer therapy (e.g., immunotherapy, chemotherapy, or biologic modifier therapy)
* Medication known to increase triglyceride levels or associated with pancreatic toxicity
* Systemic vitamin A in doses exceeding 15,000 IU/day within 14 days prior to initiating study therapy
* Concurrent gemfibrozil (Lopid^®)
* Concurrent anticancer therapy of any kind other than that mandated by the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Response rate as measured by RECIST criteria
Time to progression

SECONDARY OUTCOMES:
Survival
Patient-reported symptoms and side effects

CONTACTS AND LOCATIONS:
Overall Officials: Raghu Nandan, MD, Study Chair — Raghu Nandan, M.D., Inc
Locations (1):
- R. Nandan M.D. Incorporated, Lakewood, California, United States